CLINICAL TRIAL: NCT04010851
Title: The Effects of a Peer Co-led Educational Programme for Parents of Children With ADHD: A Feasibility Randomized Controlled Trial
Brief Title: The Effects of a Peer Co-led Educational Programme for Parents of Children With ADHD
Acronym: ADHD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: to much uncertainty about possibilities for recruiting
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Molde University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/1196/REK Mid Norway
Record Dates: First submitted 2019-06-28; First posted 2019-07-08 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Parental activation; Peer co-led education
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: The intervention is delivered in a group format, which takes the form of a full day's training, focusing on ADHD diagnosis, its treatment, how to cope with the challenges related to living with ADHD, as well as coping with challenges of parenting a child with chronic health conditions. After this one day-intervention, the participants can continue in self-help groups, which meet once a week for a 2-hour evening session. User representatives lead these weekly self-help groups, which do not require user-fees and aim to offer practical tools, support and information to increase the parent's skills, knowledge and confidence. Participants are encouraged to adopt an active role in order to achieve a positive parent/provider partnership.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer co-led educational group (Experimental): The intervention delivered in a group format is added to treatment as usual. After the parents participate in the one day-intervention, they can continue in self-help groups, which meet once a week for a 2-hour evening session. User representatives lead these weekly self-help groups, which do not require user-fees and aim to offer practical tools, support and information to increase the parent's skills, knowledge and confidence.
  Interventions: Behavioral: Peer co-led educational group
- Control group (Other): The control goup will receive treatment as usual.
  Interventions: Behavioral: Comparator treatment as usual

INTERVENTIONS:
Behavioral: Peer co-led educational group — The intervention is delivered in a group format, which takes the form of a full day's training, focusing on ADHD diagnosis, its treatment, how to cope with the challenges related to living with ADHD, as well as coping with challenges of parenting a child with chronic health conditions. After this one day-intervention, the participants can continue in self-help groups, which meet once a week for a 2-hour evening session. User representatives lead these weekly self-help groups, which do not require user-fees and aim to offer practical tools, support and information to increase the parent's skills, knowledge and confidence. Participants are encouraged to adopt an active role in order to achieve a positive parent/provider partnership.
  Arms: Peer co-led educational group
Behavioral: Comparator treatment as usual — Control group will receive treatment as usual, including different treatment options that can help alleviate the symptoms of ADHD and arm families with the tools needed to better handle problem behaviors when they arise. These interventions include: medication, psychotherapy, or a combination of these two approaches.
  Arms: Control group

SUMMARY:
ADHD is associated with a substantial burden on families, and systems pertaining to health, social care, and criminal justice, and there is a need for more knowledge of the effects of non-pharmacological interventions. Educational and parental activation interventions may improve ADHD symptoms, and may enhance parent activation. Although the results of these studies are promising, few interventions have been carried out in collaboration with user representatives, which is required by Norwegian legislation. As such, there is a need for clinical studies that document the effects of educational group interventions based on user involvement that seeks to improve parental activation. Furthermore, it is not clear which type of educational intervention that should be offered, and which aspects of parenting behaviour to focus on. There is a lack of studies investigating whether adding an intervention designed specifically for families of children with ADHD will be more effective than treatment as usual (TAU). The purpose of the present study is to determine the feasibility and expected size of a substantive randomized controlled trial comparing an ADHD peer co-led educational programme added to TAU.

DETAILED DESCRIPTION:
The primary objective of this trial is to evaluate the acceptability and feasibility of the intervention, to assure that procedures are adequate for a subsequent full size randomized controlled trial (RCT), and to determine the likely size of the trial comparing an ADHD specific parenting peer co-led intervention for parents of children with ADHD symptoms.

Specific objectives are:

(I) investigate whether parents of children recently diagnosed with ADHD are willing to be randomized to the intervention, (II) whether sufficient numbers of families can be recruited and retained such that a full-scale RCT is likely to be feasible, (III) whether research procedures and efficacy measures are feasible and acceptable to participating families and the outpatient clinics, and (IV) whether families participating in the intervention are satisfied with the intervention.

This feasibility study is not designed to detect a treatment effect, therefore a maximum of 50 parents will be recruited. The measurements will be taken in the children (at baseline and 3 months) and parents (at baseline, two weeks, pre-post intervention and 3 months follow-up) to determine the feasibility and acceptability. These measures are chosen because they address key components of the intervention (activation, quality of life and psychological well-being). Multiple measures of similar constructs will be administered where possible (e.g., psychological well-being and quality of life) to determine which measure to include in the definitive trial according to feasibility, acceptability, and sensitivity.

Feasibility assessments:

* Feasibility of recruitment.
* Acceptability of randomization and procedures will be determined by measuring loss to follow-up (post-test and 3-month follow-up), and reasons for withdrawal will be used collected.
* Acceptability of the intervention will be determined based on the number of sessions attended by participants in the peer co-led education. We will also reported on satisfaction with the program.
* Feasibility of quantitative measures will be deemed acceptable if no questionnaires are missing in full in more than 25% of the participants and if reliability was higher than 0.70.
* Follow-up response rates (post-intervention and 3 months follow-ups).

ELIGIBILITY:
Inclusion Criteria:

* Parents of children aged 6 - 12 with a formal diagnosis of ADHD, following a standardised assessment.

Exclusion Criteria:

* Participants already taking part in research on a parenting intervention will also be ineligible to participate.
* Families attending other parenting groups

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | Over a two year study period
  Feasibility of recruitment will be assessed by determining the recruitment rate, by monitoring patient screening and subsequent agreement to participate.
Satisfaction with the intervention | From baseline to 12- and 52-weeks follow-up
  Parent satisfaction will be measured by means of the client satisfaction Questionnaire, CSQ-3 as it applies to the group-based educational programme. The scale comprises three items measured on a scale from 1 (not satisfied) to 4 (very satisfied).
Parental activation | From baseline to 12- and 52-weeks follow-up
  Parental activation will be measure with the P-PAM-13. The 13-items P-PAM has four possible response options ranging from (1) strongly disagree, to (4) strongly agree, and an additional 'not applicable' option.

SECONDARY OUTCOMES:
Parental well-being | From baseline to 12- and 52-weeks follow-up
  Parental well-being will be measured by the WHO-5 Well-being Index. The questionnaire has five items rated on a six-point scale from 0 (all the time) to 5 (at no time); this items are transformed into 0-100 scales (high scores indicate a better well-being).
Parental quality of life | From baseline to 12- and 52-weeks follow-up
  Parental quality of life will be measured by the 10- items Multicultural Quality of Life Index (MQLI) which cover key aspects of the concept, from physical well-being to spiritual fulfilment. The MQLI questionnaire has ten items.
Shared decision making | From baseline to 12- and 52-weeks follow-up
  It will be assessed using a modified version of the Control Preferences Scale to provide information about the parent's preferred role in involvement.
Parental involvement in treatment decision | From baseline to 12- and 52-weeks follow-up
  Parent involvement will be assessed using a modified version of the CollaboRATE scale
Beliefs about medicines | From baseline to 12- and 52-weeks follow-up
  To investigate the beliefs about medicines we will use the Beliefs about Medicines Questionnaire (BMQ).
Adherence | From baseline to 12- and 52-weeks follow-up
  To investigate medication adherence using the Medication Adherence Rating Scale 5 items.
ADHD Scale Parent Version | From baseline to 12- and 52-weeks follow-up
  The SNAP-IV 18-Item will be use to evaluate ADHD, the SNAP-IV 18-Item Scale Parent Version is an abbreviated version of the Swanson, Nolan, and Pelham (SNAP). The questionnaire includes items for the two subsets of symptoms, inattention (items 1-9) and hyperactivity/impulsivity (items 10-18), from the DSM-IV criteria for ADHD. The scores in each of the two subsets are added together. SNAP-IV is used to measure ADHD symptoms and behavioral problems in school-aged children. Symptom severity is rated on a 4-point scale.
Level of functioning of children in Child | From baseline to 12- and 52-weeks follow-up
  The C-GAS will be used to assess the overall level of functioning of children. The C-GAS is a numeric scale ranging from 1 to 100 used to assess the overall level of functioning of children in Child and Adolescent Mental Health Services, with high scores indicating better functioning.

OTHER OUTCOMES:
Participation in treatment | From baseline to 12- and 54-weeks follow-up.
  Information regarding treatment participation and use of services will be collected via Patient Administrative System (PAS).

CONTACTS AND LOCATIONS:
Overall Officials: Ingunn P. Mundal, PhD, Principal Investigator — Molde University College; Mariela Loreto Lara Cabrera, PhD, Principal Investigator — St Olavs Hospital, Department of research and development AFFU, and NTNU; Rolf W. Gråwe, Phd prof, Study Director — Norwegian University of Science and Technology

IPD SHARING:
Plan to Share IPD: No
We anticipate that anonymised trial data may be shared with other researchers to enable international prospective meta-analyses.

REFERENCES:
- [Derived] Mundal I, Grawe RW, Hafstad H, De Las Cuevas C, Lara-Cabrera ML. Effects of a peer co-facilitated educational programme for parents of children with ADHD: a feasibility randomised controlled trial protocol. BMJ Open. 2020 Dec 2;10(12):e039852. doi: 10.1136/bmjopen-2020-039852. PMID 33268416